CLINICAL TRIAL: NCT01262248
Title: Computer-based Classification of Small Colorectal Polyps
Brief Title: Computer-based Classification of Colorectal Polyps Using Narrow-band Imaging
Status: Completed | Type: Observational
Sponsor: Tischendorf, Jens, M.D. (Individual)
Responsible Party: Tischendorf, Jens, M.D., Department of Medicine III, University of Aachen (RWTH)
Other Study IDs: Ti-NBI
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Colorectal Polyps
Keywords: small colorectal polyps; narrow band imaging; vascularization; computer-based classification
MeSH Terms: conditions — Neovascularization, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with colorectal polyps

SUMMARY:
Recent studies have shown that narrow-band imaging (NBI) is a powerful diagnostic tool for the differentiation between neoplastic and non-neoplastic colorectal polyps. The aim of the present study is to develop and evaluate a computer-based method for automated classification of small colorectal polyps on the basis of vascularization features.In a prospective study 207 polyps with a size of 10mm or smaller should be detected by a zoom NBI colonoscopy. These polyps were imaged and subsequently removed for histological analysis. the polyp images were analyzed by a computer algorithm. The proposed computer-based method consists of several steps: preprocessing, vessel segmentation, feature extraction and classification. The results of the automatic classification (sensitivity, specificity, negative predictive value, positive predictive value and accuracy)were compared to those of human observers, who were blinded to the histological gold standard.

ELIGIBILITY:
Inclusion Criteria:

* All patients who did not meet the exclusion criteria were included in the study

Exclusion Criteria:

* Patients with chronic inflammatory bowel disease, adenomatosis coli, coagulopathy, insufficient bowel preparation, or previous colonoscopy within the last 3 years; age under 18 years; no written informed consent for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent colonoscopy and colorectal polyps with a size of 10mm or smaller were detected
Sampling Method: Probability Sample
Enrollment: 434 (Actual)
Dates: Start 2010-05; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
diagnostic value (sensitivity, specificity, negative predictive value, positive predictive value, accuracy) | 10 months

SECONDARY OUTCOMES:
interobserver variability | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Jens Tischendorf, M.D., Principal Investigator — Medical Department III, University Hospital Aachen (RWTH), Pauwelsstr. 30, 52074 Aachen
Locations (1):
- Department of Medicine III, University Hospital Aachen (RWTH), Aachen, Germany

REFERENCES:
- [Background] Ignjatovic A, East JE, Suzuki N, Vance M, Guenther T, Saunders BP. Optical diagnosis of small colorectal polyps at routine colonoscopy (Detect InSpect ChAracterise Resect and Discard; DISCARD trial): a prospective cohort study. Lancet Oncol. 2009 Dec;10(12):1171-8. doi: 10.1016/S1470-2045(09)70329-8. Epub 2009 Nov 10. PMID 19910250
- [Background] Tischendorf JJ, Schirin-Sokhan R, Streetz K, Gassler N, Hecker HE, Meyer M, Tacke F, Wasmuth HE, Trautwein C, Winograd R. Value of magnifying endoscopy in classifying colorectal polyps based on vascular pattern. Endoscopy. 2010 Jan;42(1):22-7. doi: 10.1055/s-0029-1215268. Epub 2009 Nov 6. PMID 19899031